CLINICAL TRIAL: NCT02464735
Title: Effect of Sleep Disruption on the Outcome of Weaning From Mechanical Ventilation
Acronym: SLEEWE
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: REB# 15-142
Record Dates: First submitted 2015-05-28; First posted 2015-06-08 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Respiratory Insufficiency
Keywords: Sleep disruption; Spontaneous breathing trial; Weaning
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Polysomnography

SUMMARY:
Mechanically ventilated patients in the Intensive Care Unit (ICU) are highly susceptible to sleep disruption. Several studies in the last 15 years have demonstrated an extremely poor sleep quality and abnormal sleep pattern evaluated by polysomnography (PSG) devices (the gold standard method for evaluating sleep quality and quantity). Discontinuation of mechanical ventilation should be considered as soon as possible when a patient's condition starts to improve. A patient's ability to be weaned from the mechanical ventilator can be assessed using two step approaches including a Rapid Shallow Breathing Index (RSBI) calculation then a spontaneous breathing trial (SBT) to determine the likelihood of success or failure before considering endotracheal extubation. The rate of weaning failure from the first SBT attempt has been reported to be 35-55%. The reason for weaning failure may be complex and multifactorial. An association between sleep disruption and weaning outcome has never been studied. The goal of this study is to look for an association between poor sleep quality and failure of a weaning attempt.

This study is an observational, physiological study investigating sleep quality and quantity in patients who will be weaned by recording standard PSG (from 17:00 to 08:00) at night before a weaning attempt. Sleep characteristics of patients failing or passing the weaning attempt will be compared. In addition, we will compare sleep patterns before and after endotracheal extubation.

DETAILED DESCRIPTION:
This clinical physiological study will take place over a period of 2-14 days, depending on the participant.

Assessment of the readiness to wean using RSBI calculation and an SBT are standard practice in the ICU, and the decision to perform one is made by the ICU team. They are usually performed in the morning between 08:00 and 10:00. The RSBI calculation will be performed by disconnecting the patient from the ventilator for 2-3 minutes and then measuring the breathing frequency and average tidal volume for 1 minute. A value of the RSBI index < 100-105 breaths/min×L predicts a possible successful SBT. The SBT will be performed using flow-by technique (Pressure Support (PS)/Continuous Positive Airway Pressure (CPAP) 0/0 cmH2O) for 30 to 120 minutes and at a Fraction of Inspired Oxygen (FiO2) below 0.5 when the RSBI index < 100-105 breaths/min×L. A T-piece trial gives the most reliable assessment of weaning capability, but it is often reserved for the most challenging patients. Using flow-by (PS/CPAP 0/0 cmH2O) will give a similar indication of weaning capability in comparison to T-piece, but will allow the Respiratory Therapists to keep the same equipment and to monitor tidal volume and minute ventilation throughout the test. During the SBT, respiratory and hemodynamic parameters will be continuously monitored. Determining the success or failure of the SBT will be performed by the clinical team. For patients who pass the SBT, the decision for extubation is made by the ICU clinical team independently from this study. For the purpose of the study, a daily screening will be performed each afternoon by the Respiratory Therapist to identify patients who will have a RSBI calculation and an SBT the following day.

On the night prior to the planned weaning assessment, sleep architecture will be recorded using standard PSG (electroencephalography, right and left electrooculography, submental electromyography and electrocardiography) from 17:00 to 8:00. Pulse oximetry (SpO2) and end-tidal carbon dioxide (EtCO2) or transcutaneous partial pressure of carbon dioxide (PtcCO2) will be recorded continuously during the PSG.

For patients who pass the RSBI index and SBT and are extubated successfully, PSG recording will be repeated that night. If the patient passes the SBT but is not extubated, we will wait for a new extubation attempt within the next 48 hours. If extubation is performed within the next 48 hours, PSG recording will be repeated the night of extubation. If extubation is further delayed, no PSG will be performed.

For patients who fail the 1st RSBI or fail the 1st SBT, PSG recording will be repeated the night before the next weaning attempt and the night of extubation if it happens within a maximum of two weeks from the 1st SBT.

Assessment of delirium will be performed using the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) twice daily (at 08:00 and 18:00) from day 0 until extubation.

ELIGIBILITY:
Inclusion Criteria:

* Age > 16 years
* Intubated and mechanically ventilated
* A spontaneous breathing trial (SBT) is planned for the next day; patients can be enrolled if they have already had previous SBTs

Exclusion Criteria:

* Presence of recent major central nervous system disease impairing consciousness with Glasgow Coma Scale ≤ 8T
* Patients with a sleep breathing disorder when it is predominantly central sleep apnea; patients with predominantly obstructive sleep apnea can be included

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Mechanically ventilated Intensive Care Unit patients who have a spontaneous breathing trial planned for the next day.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Comparison of sleep quality between patients who pass weaning and patients who fail a weaning assessment | 15 hours
Comparison of sleep quality (sleep efficiency and fragmentation) the night before a patient fails weaning and the night after they eventually pass weaning | 30 hours

SECONDARY OUTCOMES:
Comparison between patients who pass and patients who fail weaning in terms of % of rapid eye movement sleep, sleep quantity (or efficiency), slow wave sleep and circadian sleep ratio, % of "pathological/atypical" sleep patterns, and sleep continuity | 15 hours
Comparison of sleep architecture (total sleep time, % of NREM and REM sleep) the night before weaning and the night of extubation | 30 hours
Incidence of delirium amongst all patient groups, regardless of the outcome of weaning | Up to 14 days
  Assessed using the Confusion Assessment Method for the Intensive Care Unit twice daily (at 08:00 and 18:00) each day until extubation.
Analysis of the validity of the odds ratio product (ORP) technique for classification of sleep depth in comparison to standard PSG criteria by American Academy of Sleep Medicine (AASM). | Up to 14 days
Correlation between sleep disruption and delirium. | Up to 14 days
  Assessed using the Confusion Assessment Method for the Intensive Care Unit twice daily (at 08:00 and 18:00) each day until extubation.

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - St. Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario

REFERENCES:
- [Background] Drouot X, Cabello B, d'Ortho MP, Brochard L. Sleep in the intensive care unit. Sleep Med Rev. 2008 Oct;12(5):391-403. doi: 10.1016/j.smrv.2007.11.004. Epub 2008 May 23. PMID 18502155
- [Background] Roche Campo F, Drouot X, Thille AW, Galia F, Cabello B, d'Ortho MP, Brochard L. Poor sleep quality is associated with late noninvasive ventilation failure in patients with acute hypercapnic respiratory failure. Crit Care Med. 2010 Feb;38(2):477-85. doi: 10.1097/CCM.0b013e3181bc8243. PMID 19789439
- [Background] Tobin MJ. Extubation and the myth of "minimal ventilator settings". Am J Respir Crit Care Med. 2012 Feb 15;185(4):349-50. doi: 10.1164/rccm.201201-0050ED. No abstract available. PMID 22336673
- [Background] Boles JM, Bion J, Connors A, Herridge M, Marsh B, Melot C, Pearl R, Silverman H, Stanchina M, Vieillard-Baron A, Welte T. Weaning from mechanical ventilation. Eur Respir J. 2007 May;29(5):1033-56. doi: 10.1183/09031936.00010206. PMID 17470624